# Comparison of Type 2 diabetes Pharmacotherapy Regimens Using Targeted Learning

NCT05073692

11/10/2025

# **Study Protocol**

# **Objectives**

This project aims to compare cardiovascular risks (3-point MACE) between four glucose-lowering treatment regiments (SU, DPP4, GLP1, and SGLT2) in patients with type 2 diabetes.

# Design

This project is an observational retrospective cohort study using health care data from six health care systems.

#### Methods

All study aims are addressed by estimating causal effects conceptualized by the comparisons of time-to-event outcomes between exposure regimens in ideal Randomized Clinical Trials (RCTs), i.e., RCTs with perfect compliance and no loss to follow up.

# Statistical Analysis Plan

#### **How Data Were Analyzed**

Data were analyzed using R.

# **What Statistical Methods Were Used**

We implemented Targeted Learning and Inverse Probability Weighting to estimate three classes of effect measures using longitudinal observational data: hazard ratios (HR), cumulative risk differences (RD), and differences between areas under the survival curves (also termed "restricted mean survival time"). Each of them were evaluated under both the intention-to-treat and per-protocol principles used in the analysis of RCT data.

# **How Adjustments Were Made for Covariates**

All analyses were adjusted for 400 covariates using Super Learning for propensity score estimation, and LASSO for outcome regressions.

# **Critical Assumption**

Analyses relied on the untestable no unmeasured confounding assumption.

For additional details, see:

Neugebauer R, An J, Dombrowski SK, et al. Glucose-Lowering Medication Classes and Cardiovascular Outcomes in Patients With Type 2 Diabetes. JAMA Netw Open. 2025;8(10):e2536100. doi:10.1001/jamanetworkopen.2025.36100

# **Informed Consent Form**

Not Applicable.